CLINICAL TRIAL: NCT06034483
Title: Effects of Pelvic Floor Exercise Training in Postmenopausal Genitourinary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof. Dr, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/188
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Exercise Training (Experimental): progressive pelvic floor muscle training for 8 weeks
  Interventions: Other: Pelvic floor exercise training; Other: Patient/individual education
- Patient/Individual Education (Active Comparator): Individual/patient education includes menopause, sexual health, pelvic floor health and lifestyle issues.
  Interventions: Other: Patient/individual education

INTERVENTIONS:
Other: Pelvic floor exercise training — * Pelvic floor muscle contraction will be verified with vaginal palpation and a progressive pelvic floor muscle training program will be given.
  * In the pelvic floor muscle training program:
  * Fast and slow pelvic floor muscle contractions will be taught,
  * Training will begin with 3 sets of exercises per day, exercise compliance of individuals will be monitored in the controls to be made every 2 weeks, and the number of exercise sets will be increased by one set.
  * 1 set of exercises: It will include 10 fast + 10 continuous (frequent-(3-10 sec) hold-release) contractions.
  * Individuals will be tracked with exercise diaries.
  * At the end of the 8th week, post-intervention evaluations will be made again.
  * The exercise program will be completed with a total of 6 sets of exercises per day (60 fast and 60 slow per day).
  Arms: Pelvic Floor Exercise Training
Other: Patient/individual education — In the individual/patient information training, training will be given on menopause, sexual health, pelvic floor health and lifestyle. This training will cover more specifically the following topics:
  * Explaining menopause and menopausal symptoms
  * Defining the Genitourinary Syndrome of Menopause (MGS)
  * The effect of MGS on sexual function cycle and sexual function,
  * Conservative recommendations on MGS management
  * Explaining pelvic floor anatomy and function and recommendations for pelvic floor health.
  The training will take approximately 1 hour and the training will be repeated at the end of the 1st month.

SUMMARY:
Genitourinary syndrome of menopause (MGS) is a clinical picture accompanied by genital and urinary symptoms and is commonly seen in the postmenopausal period. In the literature, the effects of drug and non-drug methods in the improvement of these symptoms have been investigated in many different designs. There is limited evidence that pelvic floor physiotherapy improves vulvovaginal blood flow with repetitive muscle activation, reduces vulvar irritation with reduction in urinary incontinence episodes, and normalizes pelvic floor muscle tone in the treatment of MGS. In addition, there is no study to the best of our knowledge investigating the effects of pelvic floor muscle exercise training and patient/individual training, in which individuals are informed. Therefore, the aim of this study is to compare the effects of pelvic floor muscle training and patient/individual information training in the presence of a physiotherapist on genitourinary symptoms and quality of life in individuals with GSM and to contribute to science in the light of this information. Before starting the study, the physical (height, body weight) and sociodemographic characteristics (age, marital status, educational status, employment status), medical history and menopausal characteristics of the individuals will be recorded. In addition, the pelvic floor muscle strength of the individuals will be evaluated at the beginning of the study and after the study is completed; genital symptoms, urinary symptoms and quality of life and scales will be questioned. Within the scope of individual/patient information education, menopause and menopause-related complaints, genitourinary (genital, sexual and urinary-related) symptoms of menopause, sexual function, the effect of menopause on sexual functions, recommendations for menopausal symptoms and complaints, and the structure and function of the pelvic floor muscles and pelvic floor muscles. Information will be given including recommendations for base health. This training will be given at the beginning of the study and will be repeated after 4 weeks to increase the benefit of the training. Individuals will be included in the progressive exercise training program within the scope of the pelvic floor muscle exercise training program. In the controls to be made every 15 days, the exercise compliance of the individuals will be monitored and the number of exercises will be increased. Exercise charts will be given in order to increase the adaptation of individuals to exercise and the benefit they will gain from exercise. The estimated time in this study is 8 weeks and it is planned to include 50 volunteers in the study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study and signing the informed consent form,
* Being between the ages of 40-75
* Being in the postmenopausal period (last menstrual period >12 months ago),
* Having at least 1 genital (vaginal dryness, dyspareunia, vulvovaginal itching/irritation, etc.) and urinary symptoms (dysuria, urinary incontinence, etc.),
* Active pelvic floor muscle contraction ability,
* Absence of any mental problem/cooperation problem that prevents completing the study scales.

Exclusion Criteria:

* Presence of vulvo-vaginal dermatological diseases or neoplasia,
* a history of pelvic organ cancer,
* pelvic radiation exposure,
* signs of vaginal or urinary infection,
* history of medical or surgical treatment for urinary incontinence (eg, mid-urethral sling, pubovaginal sling)
* history of pelvic surgery (hysterectomy, pelvic prolapse surgery, etc.)
* presence of advanced pelvic organ prolapse (prolapse stage >stage 2 according to the pelvic organ prolapse staging system),
* presence of morbid obesity (body mass index ≥35 kg/m2),
* the presence of cognitive disorders and neuropsychiatric diseases (Alzheimer's, dementia, Parkinson's, etc.),
* use of antiestrogenic drugs,
* taking hormone replacement therapy

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
vulvovaginal symptoms | change in severity of vulvovaginal symptoms from baseline up to end of 8th weeks
  Vulvovaginal Symptom Questionnaire will be used to evaluate vulvovaginal symptoms severity . This questionnaire consists of three parts. The first two sections are answered by all women, regardless of current sexual activity. The first 7 questions of the questionnaire include the symptom subscale and in the last week; It includes questions about itching, burning, soreness, irritation, dryness, discharge and odor. The next section of the VSQ assesses the emotional and lifestyle impact of vulvovaginal symptoms during the past week. In the third part, the effect of vulvovaginal symptoms on sexual function in sexually active women is questioned.
urinary symptoms | change in severity of urinary symptoms from baseline up to end of 8th weeks
  International consultation on incontinence questionnaire short form will be used to evaluate urinary symptoms. This scale, which measures the severity of urinary incontinence and its effect on quality of life, has four sub-dimensions. In the first dimension, the frequency of urinary incontinence, the amount of urinary incontinence in the second dimension, the effects of urinary incontinence on daily life in the third dimension, and the situations that cause urinary incontinence in the fourth dimension are questioned. The first three dimensions are scored in the evaluation.

SECONDARY OUTCOMES:
Pelvic floor muscle function and strength | change in pelvic floor muscle strength from baseline to end of 8th weeks
  Urinary stop test will be used to question the individual's ability to stop voiding during voiding and to obtain information about the strength of the pelvic floor.
Pelvic floor muscle strength | change in pelvic floor muscle strength from baseline to end of 8th weeks
  Digital palpation will be used to obtain information about the person's pelvic floor muscle strength.In digital palpation, the therapist gently inserts index and middle fingers into the vagina, a natural opening of the body, wearing a sterile glove and using lubricating gel. The patient is asked to squeeze the therapist's fingers as hard as possible. This method is a painless, easy and practical method for the evaluation of pelvic floor muscle function. It is a basic assessment method for performing exercises correctly. The strength of the contraction felt around the finger is scored according to the Modified Oxford Scale. This six-point scale is graded as 0: No contraction, 1: Vibration, 2: Weak, 3: Moderate, 4: Good, 5: Strong.
The daily effect of vaginal aging | change in the effects of menopause specific vaginal symptoms over the last 4 weeks from baseline to the 8th weeks
  The Day-to-Day impact of vaginal aging questionnaire (DIVA) will be used to evaluate the effects of menopause-specific vaginal symptoms over the last 4 weeks. The questionnaire evaluates daily life activity, emotional/behavioral status, sexual function and self-perception/body image as versatile with 4 sub-headings and 22 Likert-type questions. Each item is scored between 0-4 (0=not at all, 1=somewhat, 2=moderate, 3=quite, and 4=a lot). Higher scores indicate a higher impact of vaginal symptoms.
Urinary symptoms | change in degree of discomfort associated with urinary symptoms from baseline to end of 8th weeks
  The urinary distress inventory will be used to evaluate the urinary symptoms associated with pelvic floor dysfunction and the degree of discomfort associated with these symptoms. The best score is 0, the worst score is 100. In other words, the higher the score, the higher the level of discomfort.
Quality of life assessment | change in quality of life in postmenopausal period from baseline to end of 8th weeks
  Menopause-specific quality of life(The MENQOL) will be used to evaluate the quality of life of individuals in the menopausal period. This scale consists of four sub-dimensions, namely vasomotor, psychosocial, physical and sexual dimensions, and 32 questions. The score of each sub-dimension ranges from 1 to 8, and an increase in the score means that the relevant sub-dimension is more affected.

CONTACTS AND LOCATIONS:
Locations (1):
- Gizem Taşkıran, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercier J, Morin M, Zaki D, Reichetzer B, Lemieux MC, Khalife S, Dumoulin C. Pelvic floor muscle training as a treatment for genitourinary syndrome of menopause: A single-arm feasibility study. Maturitas. 2019 Jul;125:57-62. doi: 10.1016/j.maturitas.2019.03.002. Epub 2019 Mar 29. PMID 31133219
- [Background] Mercier J, Morin M, Tang A, Reichetzer B, Lemieux MC, Samir K, Zaki D, Gougeon F, Dumoulin C. Pelvic floor muscle training: mechanisms of action for the improvement of genitourinary syndrome of menopause. Climacteric. 2020 Oct;23(5):468-473. doi: 10.1080/13697137.2020.1724942. Epub 2020 Feb 27. PMID 32105155
- [Background] Mercier J, Morin M, Lemieux MC, Reichetzer B, Khalife S, Dumoulin C. Pelvic floor muscles training to reduce symptoms and signs of vulvovaginal atrophy: a case study. Menopause. 2016 Jul;23(7):816-20. doi: 10.1097/GME.0000000000000620. PMID 27219835